CLINICAL TRIAL: NCT04908475
Title: A Phase 4 Multicenter, Randomized, Open-label, Efficacy Assessor-blinded Study of Risankizumab Compared to Apremilast for the Treatment of Adult Subjects With Moderate Plaque Psoriasis Who Are Candidates for Systemic Therapy
Brief Title: Study of Subcutaneous Risankizumab Injection Compared to Oral Apremilast Tablets to Assess Change in Disease Activity And Adverse Events in Adult Participants With Moderate Plaque Psoriasis Who Are Candidates for Systemic Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M20-326; 2020-005512-21 (EudraCT Number)
Record Dates: First submitted 2021-05-28; First posted 2021-06-01 (Actual); Results first posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Psoriasis
Keywords: Psoriasis; Plaque Psoriasis; Risankizumab; ABBV-066; Skyrizi; Apremilast
MeSH Terms: conditions — Psoriasis | interventions — risankizumab; apremilast

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Risankizumab (Experimental): Risankizumab 150 mg as a single subcutaneous (SC) injection at at Baseline (Day 1) and Week 4 (Period A) and at Weeks 16, 28, and 40 (Period B).
  Interventions: Drug: Risankizumab
- Apremilast (Experimental): Participants receive apremilast 30 mg orally twice daily (BID) in Period A and re-randomized to receive either risankizumab 150 mg as a single SC injection at Weeks 16, 20, 32 in Period B or apremilast 30 mg orally BID from Week 16 up to Week 52 in Period B. For those taking apremilast in Period B, non-responders at Week 28 and Week 40 will be offered to receive risankizumab as rescue medication.
  Interventions: Drug: Risankizumab; Drug: Apremilast

INTERVENTIONS:
Drug: Risankizumab — Subcutaneous injection
  Other Names: ABBV-066; Skyrizi
Drug: Apremilast — Oral Tablets
  Other Names: Otezla
  Arms: Apremilast

SUMMARY:
Psoriasis (PsO) is a chronic disease characterized by marked inflammation of the skin that results in thick, red, scaly plaques. This study will assess how safe and effective risankizumab is compared to apremilast in adult participants with moderate plaque psoriasis. Adverse events and change in disease symptoms will be monitored.

Risankizumab (Skyrizi) and apremilast are approved drugs for the treatment of moderate to severe PsO. Approximately 330 participants with moderate plaque psoriasis (PsO) will be enrolled across approximately 55 sites globally.

The study has 2 periods : Period A from Baseline to Week 16, and Period B, from Week 16 to Week 52. In Period A, participants will be randomly placed into 2 groups to receive either subcutaneous risankizumab or oral apremilast for 16 weeks. In Period B, participants who received apremilast in Period A will again be randomly assigned to 1 of the 2 groups to receive either risankizumab or apremilast for 36 weeks. At weeks 28 and 40, participants considered non-responders to apremilast based on their psoriasis score will be offered to receive risankizumab.

There may be a higher burden for participants in this study compared to usual standard of care. Participants will attend regular visits per routine clinical practice. The effect of the treatment will be checked by medical assessments, checking for side effects, and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

- Candidates for systemic therapy with moderate chronic plaque psoriasis (PsO) (with or without psoriatic arthritis) at Screening and Baseline for at least 6 months prior to Baseline defined as:

* Body Surface Area (BSA) >= 10% and <= 15%; and
* Psoriasis Area and Severity Index (PASI) >= 12; and
* Static Physician Global Assessment (sPGA) = 3 (moderate) based on a 5-point scale (0 to 4).

Exclusion Criteria:

* Participant has any form of PsO other than chronic plaque PsO (e.g., pustular PsO, palmoplantar pustulosis, acrodermatitis of Hallopeau, erythrodermic, or guttate PsO).
* History of current drug-induced PsO or a drug-induced exacerbation of pre-existing psoriasis.
* History of active ongoing inflammatory skin diseases other than PsO and psoriatic arthritis that could interfere with the assessment of PsO (e.g., hyperkeratotic eczema).
* Prior exposure to risankizumab or apremilast.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (54):
- United States (26):
  - Total Skin and Beauty Dermatology Center /ID# 233793, Birmingham, Alabama
  - Advanced Research Associates - Glendale /ID# 229266, Glendale, Arizona
  - Alliance Dermatology and MOHs Center, PC /ID# 229224, Phoenix, Arizona
  - UC Davis Health /ID# 229133, Sacramento, California
  - Florida Academic Centers Research and Education /ID# 229235, Coral Gables, Florida
  - Olympian Clinical Research - Largo /ID# 233792, Largo, Florida
  - Renstar Medical Research /ID# 228946, Ocala, Florida
  - ForCare Clinical Research /ID# 229135, Tampa, Florida
  - Arlington Dermatology /ID# 228945, Rolling Meadows, Illinois
  - Dawes Fretzin, LLC /ID# 229010, Indianapolis, Indiana
  - Epiphany Dermatology of Kansas LLC /ID# 229221, Overland Park, Kansas
  - DermAssociates, LLC /ID# 229016, Rockville, Maryland
  - Michigan Center for Research Company /ID# 229136, Clarkston, Michigan
  - Henry Ford Medical Center /ID# 229215, Detroit, Michigan
  - MediSearch Clinical Trials /ID# 229269, Saint Joseph, Missouri
  - Physician Research Collaboration, LLC /ID# 229225, Lincoln, Nebraska
  - Advanced Dermatology of the Midlands /ID# 229009, Omaha, Nebraska
  - Psoriasis Treatment Center of Central New Jersey /ID# 228943, East Windsor, New Jersey
  - University Hospitals Case Medical Center /ID# 229240, Cleveland, Ohio
  - Wright State Physicians - Fairborn /ID# 230051, Fairborn, Ohio
  - Oregon Dermatology and Research Center /ID# 233462, Portland, Oregon
  - Arlington Research Center, Inc /ID# 229264, Arlington, Texas
  - Bellaire Dermatology Associates /ID# 230118, Bellaire, Texas
  - Center for Clinical Studies - Houston (Binz) /ID# 229263, Houston, Texas
  - Center for Clinical Studies - Houston (Binz) /ID# 229272, Houston, Texas
  - Premier Clinical Research /ID# 229220, Spokane, Washington
- Canada (9):
  - Beacon Dermatology Inc /ID# 230121, Calgary, Alberta
  - Dr. Chih-ho Hong Medical Inc. /ID# 230337, Surrey, British Columbia
  - Enverus Medical Research /ID# 230480, Surrey, British Columbia
  - Karma Clinical Trials /ID# 230339, St. John's, Newfoundland and Labrador
  - Dermatrials Research /ID# 230119, Hamilton, Ontario
  - Dr. S.K. Siddha Medicine Professional Corporation /ID# 230416, Newmarket, Ontario
  - K. Papp Clinical Research /ID# 230336, Waterloo, Ontario
  - Innovaderm Research Inc. /ID# 230334, Montreal, Quebec
  - Centre de Recherche dermatologique du Quebec Metropolitain /ID# 230478, Québec, Quebec
- Germany (9):
  - Universitaetsklinikum Erlangen /ID# 229433, Erlangen, Bavaria
  - Universitaetsklinikum Frankfurt /ID# 229431, Frankfurt am Main, Hesse
  - Universitaetsklinikum Muenster /ID# 229432, Munster, Lower Saxony
  - DermaKiel Allergie und Haut Centrum /ID# 229630, Kiel, Schleswig-Holstein
  - Fachklinik Bad Bentheim /ID# 231504, Bad Bentheim
  - Hautarztpraxis Dr. Niesmann und Dr. Othlinghaus /ID# 230245, Bochum
  - SRH Wald-Klinikum Gera /ID# 229445, Gera
  - MENSINGDERMA research GmbH /ID# 229435, Hamburg
  - Dermatologische Gemeinschaftspraxis Mahlow /ID# 229434, Mahlow
- Israel (4):
  - Rambam Health Care Campus /ID# 229620, Haifa, H_efa
  - Rabin Medical Center /ID# 229074, Haifa, H_efa
  - HaEmek Medical Center /ID# 231901, Afula, Southern District
  - The Chaim Sheba Medical Center /ID# 229075, Ramat Gan, Tel Aviv
- Poland (6):
  - High-Med Przychodnia Specjalistyczna /ID# 229023, Warsaw, Masovian Voivodeship
  - Royalderm Agnieszka Nawrocka /ID# 228973, Warsaw, Masovian Voivodeship
  - Uniwersytecki Szpital Kliniczny im. F. Chopina w Rzeszowie /ID# 229022, Rzeszów, Podkarpackie Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o. /ID# 229053, Gdansk, Pomeranian Voivodeship
  - Centrum Kliniczno-Badawcze J.Brzezicki, B. Gornikiewicz-Brzezicka Lekarze Spolka /ID# 228971, Elblag, Warmian-Masurian Voivodeship
  - Dermed Centrum Medyczne Sp. z o.o /ID# 229051, Lodz, Łódź Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Stein Gold LF, Bagel J, Tyring SK, Hong HC, Pavlovsky L, Vender R, Pinter A, Reich A, Drogaris L, Wu T, Patel M, Soliman AM, Photowala H, Stakias V, Richter S, Papp KA. Comparison of risankizumab and apremilast for the treatment of adults with moderate plaque psoriasis eligible for systemic therapy: results from a randomized, open-label, assessor-blinded phase IV study (IMMpulse). Br J Dermatol. 2023 Oct 25;189(5):540-552. doi: 10.1093/bjd/ljad252. PMID 37488811
- See also: Related Info — https://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 352 participants were enrolled from 48 sites across 5 countries including Canada, Germany, Israel, Poland, and the United States.
Pre-assignment Details: Period A: participants were randomized in a 1:2 ratio to risankizumab (RZB) or apremilast (APR). Period B: participants receiving RZB were continued up to Week 52; participants receiving APR were re-randomized in a 1:1 ratio to receive either RZB or APR (with the option to receive RZB as rescue) up to Week 52. Rerandomization was stratified by Psoriasis Area and Severity Index (PASI) 75 response (responder, non-responder) at Week 16.
Groups:
- Period A: APR: Apremilast 30 mg orally twice daily (BID) up to Week 16
- Periods A/B: RZB/RZB: Risankizumab 150 mg as a single subcutaneous (SC) injection at Baseline (Day 1) and Week 4 (Period A) and at Weeks 16, 28, and 40 (Period B).
- Period B: APR/APR, NR: Participants who were randomized to apremilast in Period A, failed to achieve PASI 75 at Week 16 (non-responders [NR]) and were re-randomized to apremilast 30 mg orally BID up to Week 52.
- Period B: APR/RZB, NR: Participants who were randomized to apremilast in Period A, failed to achieve PASI 75 at Week 16 (NR) and were re-randomized to risankizumab 150 mg as a single SC injection at Weeks 16, 20, 32, and 44.
- Period B: APR/APR, R: Participants who were randomized to apremilast in Period A, achieved PASI 75 at Week 16 (responders [R]) and were re-randomized to apremilast 30 mg orally BID up to Week 52.
- Period B: APR/RZB, R: Participants who were randomized to apremilast in Period A, achieved PASI 75 at Week 16 (R) and were re-randomized to risankizumab 150 mg as a single SC injection at Weeks 16, 20, 32, and 44.
Period: Period A (Baseline to Week 16)
Arm/Group | Period A: APR | Periods A/B: RZB/RZB | Period B: APR/APR, NR | Period B: APR/RZB, NR | Period B: APR/APR, R | Period B: APR/RZB, R
Started | 234 | 118 | 0 | 0 | 0 | 0
Completed | 216 | 118 | 0 | 0 | 0 | 0
Not Completed | 18 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 0 | 0 | 0 | 0 | 0
Not completed — Other, Not Specified | 6 | 0 | 0 | 0 | 0 | 0
Period: Period B (Week 16 to Week 52)
Arm/Group | Period A: APR | Periods A/B: RZB/RZB | Period B: APR/APR, NR | Period B: APR/RZB, NR | Period B: APR/APR, R | Period B: APR/RZB, R
Started (Participants re-randomized in Period B) | 0 | 118 | 78 | 83 | 22 | 20
Received ≥ 1 Dose of Study Drug | 0 | 116 | 75 | 82 | 22 | 20
Received RZB as Rescue Medication | 0 | 0 | 47 | 0 | 1 | 0
Completed | 0 | 69 | 42 | 57 | 15 | 13
Not Completed | 0 | 49 | 36 | 26 | 7 | 7
Not completed — Lost to Follow-up | 0 | 6 | 4 | 6 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 5 | 13 | 2 | 3 | 0
Not completed — Other, Not Specified | 0 | 38 | 19 | 18 | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Period A: APR: Apremilast 30 mg orally BID up to Week 16
- Period A: RZB: Risankizumab 150 mg as a single SC injection at Baseline (Day 1) and Week 4.
- Total: Total of all reporting groups
Arm/Group | Period A: APR | Period A: RZB | Total
Number analyzed (Participants) | 234 | 118 | 352
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (14.27) | 45.5 (13.63) | 46.0 (14.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 42 | 121
  Male | 155 | 76 | 231
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 7 | 30
  Not Hispanic or Latino | 211 | 111 | 322
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 14 | 12 | 26
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 9 | 5 | 14
  White | 209 | 98 | 307
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Psoriasis Area Severity Index (PASI) 90 (Defined as at Least 90% Improvement in PASI From Baseline) in Intent to Treat Population at Week 16 (ITT_A)
Description: The PASI is used to evaluate a participant's overall psoriasis disease state that includes the percent of surface area of skin that is affected and the severity of erythema, induration, and desquamation over four body regions (head, upper extremities, trunk, and lower extremities). Scores range from 0 to 72, with higher scores indicating more severe disease.
Time Frame: Week 16
Population: ITT_A Population: all participants randomized in Period A
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Period A: APR | Period A: RZB
Number analyzed (Participants) | 234 | 118
percentage of participants | 5.1 [2.3 to 8.0] | 55.9 [47.0 to 64.9]
Statistical Analysis 1: Comparison: Period A: APR vs Period A: RZB; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Adjusted for strata (baseline body weight [≤ 100 kg, > 100 kg] and prior exposure to any systemic and/or biologic treatment for psoriasis [0, ≥ 1]) for the comparison of 2 treatment groups; Adjusted Difference = 50.7, 95% CI 2-sided [41.3 to 60.1]

2. Primary Outcome: Percentage of Participants Achieving Static Physician Global Assessment (sPGA) 0 or 1 With at Least 2-grade Improvement From Baseline in Intent to Treat Population at Week 16 (ITT_A)
Description: The sPGA is the physician's current assessment of the average thickness, erythema, and scaling of all psoriatic lesions. Scores range from 0 (clear) to 4 (severe).
Time Frame: Week 16
Population: ITT_A Population: all participants randomized in Period A.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Period A: APR | Period A: RZB
Number analyzed (Participants) | 234 | 118
percentage of participants | 18.4 [13.4 to 23.3] | 75.4 [67.7 to 83.2]
Statistical Analysis 1: Comparison: Period A: APR vs Period A: RZB; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted Difference = 56.8, 95% CI 2-sided [47.7 to 66.0]

3. Primary Outcome: Percentage of Participants Achieving PASI 90 in Intent to Treat Population for Apremilast Non-Responders at Week 52 (ITT_B_NR)
Description: as for outcome 1
Time Frame: Week 52
Population: ITT_B_NR Population: participants randomized to APR at Baseline who failed to achieve PASI 75 at Week 16 and were re-randomized to APR or RZB in Period B.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Period B: APR/APR, NR | Period B: APR/RZB, NR
Number analyzed (Participants) | 78 | 83
percentage of participants | 2.6 [0.0 to 6.1] | 72.3 [62.7 to 81.9]
Statistical Analysis 1: Comparison: Period B: APR/APR, NR vs Period B: APR/RZB, NR; Test type: Superiority; p < 0.001, Chi-squared; Difference = 69.7, 95% CI 2-sided [59.5 to 80.0]

4. Secondary Outcome: Percentage of Participants Achieving PASI 75 (Defined as at Least 75% Improvement in PASI From Baseline) in Intent to Treat Population at Week 16 (ITT_A)
Description: as for outcome 1
Time Frame: Week 16
Population: ITT_A Population: all participants randomized in Period A
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Period A: APR | Period A: RZB
Number analyzed (Participants) | 234 | 118
percentage of participants | 18.8 [13.8 to 23.8] | 84.7 [78.3 to 91.2]
Statistical Analysis 1: Comparison: Period A: APR vs Period A: RZB; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Adjusted for strata (baseline body weight [≤ 100 kg, > 100 kg] and prior exposure to any systemic and/or biologic treatment for psoriasis [0, ≥ 1] for the comparison of 2 treatment groups; Adjusted Difference = 65.9, 95% CI 2-sided [57.6 to 73.9]

5. Secondary Outcome: Percentage of Participants Achieving PASI 75 in Intent to Treat Population for Apremilast Non-Responders at Week 52 (ITT_B_NR)
Description: as for outcome 1
Time Frame: Week 52
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Period B: APR/APR, NR | Period B: APR/RZB, NR
Number analyzed (Participants) | 78 | 83
percentage of participants | 11.5 [4.4 to 18.6] | 83.1 [75.1 to 91.2]
Statistical Analysis 1: Comparison: Period B: APR/APR, NR vs Period B: APR/RZB, NR; Test type: Superiority; p < 0.001, Chi-squared; Difference = 71.6, 95% CI 2-sided [60.9 to 82.3]

6. Secondary Outcome: Percentage of Participants Achieving Static Physician Global Assessment (sPGA) 0 or 1 With at Least 2-grade Improvement From Baseline in Intent to Treat Population for Apremilast Non-Responders at Week 52 (ITT_B_NR)
Description: as for outcome 2
Time Frame: Week 52
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Period B: APR/APR, NR | Period B: APR/RZB, NR
Number analyzed (Participants) | 78 | 83
percentage of participants | 7.7 [1.8 to 13.6] | 77.1 [68.1 to 86.1]
Statistical Analysis 1: Comparison: Period B: APR/APR, NR vs Period B: APR/RZB, NR; Test type: Superiority; p < 0.001, Chi-squared; Difference = 69.4, 95% CI 2-sided [58.6 to 80.2]

ADVERSE EVENTS:
Time Frame: All Cause Mortality: From enrollment up to end of study, for an overall median of 419.5 days. Adverse Events: From first dose of study drug through approximately 20 weeks (140 days) after administration of the last dose of RZB (i.e., Week 40 for participants originally randomized to RZB and Week 44 for participants switched from APR to RZB) or approximately 4 weeks (28 days) after the last dose of APR (i.e., Week 56 for participants who remain on the APR arm after re-randomization).
Description: Safety Population: participants who received ≥ 1 dose of study drug. Note: Response at Week 16 was not applicable to the Safety Reporting Groups.
Groups:
- Period A: RZB: Risankizumab 150 mg as a single SC injection at Day 1 and Week 4
- Period B: RZB/RZB: Participants who received risankizumab 150 mg as a single subcutaneous (SC) injection at Day 1 and continued on risankizumab at Weeks 16, 28, and 40
- Period B: APR/APR: Participants who received apremilast in Period A who were re-randomized to receive apremilast 30 mg orally BID up to Week 52.
- Period B: APR/RZB: Participants who received apremilast in Period A who were re-randomized to receive risankizumab 150 mg as a single SC injection at Weeks 16, 20, 32, 44.
- Period B: APR/APR/RZB: Participants who received apremilast in Period A who were re-randomized to receive apremilast 30 mg orally BID and received rescue medication with risankizumab.
Arm/Group | Period A: APR | Period A: RZB | Period B: RZB/RZB | Period B: APR/APR | Period B: APR/RZB | Period B: APR/APR/RZB
All-Cause Mortality (participants affected / at risk) | 0/234 | 0/118 | 0/116 | 0/97 | 0/102 | 0/48
Serious Adverse Events (participants affected / at risk) | 4/234 | 1/118 | 8/116 | 2/97 | 3/102 | 0/48
Other Adverse Events (participants affected / at risk) | 101/234 | 24/118 | 36/116 | 27/97 | 31/102 | 15/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period A: APR (N=234) | Period A: RZB (N=118) | Period B: RZB/RZB (N=116) | Period B: APR/APR (N=97) | Period B: APR/RZB (N=102) | Period B: APR/APR/RZB (N=48)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OBSTRUCTIVE PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
UMBILICAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
APPENDICITIS PERFORATED (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OSTEOCHONDROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CAROTID ARTERY STENOSIS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GENERALISED TONIC-CLONIC SEIZURE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SCIATICA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NASAL INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period A: APR (N=234) | Period A: RZB (N=118) | Period B: RZB/RZB (N=116) | Period B: APR/APR (N=97) | Period B: APR/RZB (N=102) | Period B: APR/APR/RZB (N=48)
DIARRHOEA (Gastrointestinal disorders) | 47 (50) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 41 (45) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 16 (16) | 13 (13) | 19 (20) | 14 (14) | 12 (12) | 6 (6)
NASOPHARYNGITIS (Infections and infestations) | 10 (13) | 4 (5) | 11 (14) | 8 (10) | 10 (11) | 5 (6)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 3 (3) | 5 (5) | 3 (3) | 6 (8) | 1 (1)
HEADACHE (Nervous system disorders) | 27 (28) | 3 (3) | 1 (1) | 4 (4) | 5 (6) | 1 (1)
HYPERTENSION (Vascular disorders) | 3 (3) | 2 (2) | 6 (6) | 0 (0) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/75/NCT04908475/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-26): https://cdn.clinicaltrials.gov/large-docs/75/NCT04908475/SAP_001.pdf